CLINICAL TRIAL: NCT01013298
Title: Video-guided Percutaneous Tracheostomy (PCT): Evaluating the Safety, Efficacy and Simplicity of a Novel Technique
Brief Title: Video-guided Percutaneous Tracheostomy (PCT): A Feasibility Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Prof Patrick Sorkine, Intensive Care unit, Tel aviv Sourasky Medical center
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Supportive Care
Other Study IDs: TASMC-09-PS-0543-CTIL
Record Dates: First submitted 2009-11-11; First posted 2009-11-13 (Estimated); Last update posted 2009-11-13 (Estimated); Status verified 2009-11

CONDITIONS: Bleeding; Hypoxia; Atelectasis; Pneumothorax; Pneumomediastinum
Keywords: percutaneous tracheostomy; paratracheal insertion; tracheal injury; transtracheal needle; ventilatory parameters
MeSH Terms: conditions — Hemorrhage; Hypoxia; Pulmonary Atelectasis; Pneumothorax; Mediastinal Emphysema

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- Video-guided PCT (Experimental): Patients that will be extubated and re-intubated with the ETT-TVT, and monitored throughout intubation and PCT
  Interventions: Device: video-guided PCT

INTERVENTIONS:
Device: video-guided PCT — extubation and then re-intubation with the ETT-TVT, followed by video monitoring of the PCT procedure via the ETT-TVT
  Other Names: monitored PCT

SUMMARY:
The purpose of this study is to determine the feasibility, safety and effectiveness of an endotracheal tube embedded with a mini video-camera as a guiding tool for percutaneous tracheostomy.

DETAILED DESCRIPTION:
Background

Percutaneous tracheostomy (PCT) is commonly used in the intensive care unit (ICU) for critically-ill patients who require long-term mechanical ventilation. In experienced hands, and with proper patient selection, it is safe, easy and quick, and the associated perioperative complication rate can be reduced to approximately 4% [1-7]. However, skilled intensivist may not always be available, and the procedure may sometimes entail complications. These include paratracheal insertion of the tracheostomy tube, tracheal injury; puncturing the cuff and transfixing the endotracheal tube (ETT) during the transtracheal needle insertion; inserting the guide wire through Murphy's eye; or accidental extubation while withdrawing the endotracheal tube during the procedure leading to loss of the airway [8-13].

Although using the fingertip to palpate the trachea and endotracheal tube is a useful technique to locate the tip of the endotracheal tube during the procedure, it is unreliable, particularly in patients with short and thick necks. Bronchoscopic guidance of PCT is generally recommended to minimize the risk of unintentional tracheal injury. The use of a fibreoptic bronchoscope may be helpful [14-18]. However, it is an expensive tool which is not readily available in some centers. Video guidance provides a cost-effective alternative to bronchoscopes, that may also reduce the risk of procedure-related complications such as paratracheal insertion of the tracheostomy tube, tracheal injury or cuff puncture [19].

The goal of this study is to observe and describe a simple and safe technique - Video-guided PCT - that may overcome some of the limitations of percutaneous tracheostomy, to report any potentially-related complications that may occur during or after the procedure, and to portray a learning curve obtained with this technique.

The equipment used for this technique is the ETView TVTTM, a commercially available ETT, embedded with a mini video-camera at the tip of the tube. It provides direct endoscopic visualization of the larynx and tracheal mucosa, and thereafter allows the determination of the tip of the transtracheal needle during percutaneous puncture of the trachea, and hence may reduce the likelihood of paratracheal insertion, tracheal injury, or other technical complications.

The ETView TVTTM device is compatible with any medical grade NTSC video monitor, thereby it provides monitoring of the airways during the intubation and PCT procedure, as well as continuous viewing of the airways as long as mechanical ventilation is required (www.etview.com).

Study Objectives

To observe a new bedside technique of video-guided PCT, to report any potentially-related complications, and to construct learning curves based on the operative time and complication rate.

Study design

The study will be conducted as a prospective observational one. The setting will be the ICU of the Sourasky medical center. 10 consecutive adult critically ill patients who require elective tracheostomy will be recruited for the study. Informed consent will be obtained from the families or next of kin of all study patients. In the absence of relatives, consent will be given by an anesthesiologist/intensivist not related to the study. The procedure will be performed by the same team of intensivists upon all study patients. During and following the procedure we will assess the complication rate, operative time, and operability of the procedure (see "procedure & follow-up" section).

Methods

The procedure

The procedure will be performed by an ICU team which includes: an anesthesiologist/intensivist who executes the procedure, another anesthesiologist who applies anesthetics & analgesia, a nurse, and a forth person who takes time.

During the procedures oxygen saturation, end tidal carbon dioxide (ETCO2), ECG, blood pressure, and arterial blood gases will be monitored continuously.

The video-guided PCT procedure requires extubation and re-intubation with the TVTTM tube, which will be mentioned in the consent form.

Re-intubation with the TVTTM tube will be performed as any commonly practiced intubation.

The ETView Tracheoscopic system (TVTTM) consists of an ETT, embedded with a video imaging device and a light source at its tip and an integrated cable with a connector, that may be wired to any video monitor.

The imaging system will be used to monitor the airways while intubating and, beyond the vocal cords, to locate the transtracheal insertion site and needle. In addition, the light source will serve for transillumination of the neck soft tissues, in order to delineate the tracheal curvature and identify anatomical deviations.

Anesthesia and analgesia will be routinely performed, and standardized for all the study patients. Low doses of the opiate fentanyl (2-3 μg/kg) and the short-acting sedative propofol (20 mg bolus, and 3-6mg/kg/h drip) will be administered at the beginning of the procedure. Rocuronium bromide, a brief acting muscle paralyzer, 0.6mg/kg, will also be used in most patients.

Patient follow-up

The executing physician will answer a questionnaire evaluating the intraprocedural difficulties, complications, feasibility, confidence, and operability, and will follow-up the patients during the first 6h after the procedure, or until discharge. Follow-up will include documentation of any procedure-related complications, monitoring of respiratory/ventilatory parameters and length of stay (LOS) in the ICU beyond 6h (due to medical circumstances related to the procedure).

All study patients will be placed with arterial lines through which we withdraw blood before and after the procedure, and when indicated by deterioration of respiratory parameters - for blood gas analyses (PaO2/FiO2, PaCO2, pH and BE). In addition, saturation will be documented hourly. All patients will also have chest x-rays performed immediately following tracheostomy.

The questionnaire will include a check-list listing procedure-related complications, through which we will evaluate the total number of complications. These include:

A. Technical complications: False route/paratracheal insertion, injury to a thoracic vessel, tracheal/laryngeal/esophageal injury, accidental decannulation, puncturing the cuff, inserting the guide wire through Murphy's eye, malpositioning or kinking of the tracheal cannula, failed trachestomy, multiple punctures (≥3).

B. Clinical complications potentially related to the procedure:

B.1. Intraprocedural: significant endotracheal bleeding and transfusion requirements (RBC, FFP or platelets), transient hypoxia/hypoxemia, hemodynamic changes (e.g., transient hypotension not related to anesthetics).

B.2. Postprocedure: alterations in respiratory function (defined as >15% reduction in saturation or PaO2/FiO2, compared to baseline; Increased PaCO2 without change in saturation; the need to change ventilatory settings and/or add PEEP within the first 24 hrs), atelectasis, pneumothorax, pneumomediastinum, aspiration, early unexplained mortality (within the first 24 hrs).

Other parameters they will be asked to evaluate will be: whether the transtracheal needle was recognized via the TVTTM (yes/no); intraoperative difficulties; level of confidence; ease of performance ("best practice"); and need to convert to surgical tracheostomy procedure.

In addition, a member of the team will measure operative time, which includes the total duration of the procedure; the time it took to recognize the tracheal insertion site and needle; and the time since ETT placement and until successful tracheal placement is confirmed via air bubbles or ETCO2.

The complication rate and operative time will be used to construct a learning curve for the executing intensivist.

ELIGIBILITY:
Inclusion Criteria:

* The investigators will enroll for this study
* patients aged > 18 years old, admitted to the ICU,
* who require elective PCT for prolonged mechanical ventilation, airway protection or weaning failure.

Exclusion Criteria:

* Patients indicated for surgical tracheostomy, due to altered or difficult local anatomy;
* necessity of emergency airway access due to acute airway compromise;
* evidence of infection in the soft tissues of the neck;
* coagulation abnormalities (INR>1.5, PTT>40, thrombocyte count < 50,000);
* gross distortion of the neck anatomy (due to hematoma/tumor/thyromegaly/scarring from previous neck surgery/ unstable C-spine);
* contra-indication for re-intubation/suspected loss of airway during re-intubation;
* hemodynamic instability.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2010-01; Primary Completion 2010-06 (Estimated); Study Completion 2010-08 (Estimated)

PRIMARY OUTCOMES:
procedure-related complications | 6h

SECONDARY OUTCOMES:
operative time | minutes

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Sorkine, MD, Study Director — Tel-Aviv Sourasky Medical Center; Idit Matot, MD, Study Chair — Tel-Aviv Sourasky Medical Center; Dima Shmain, MD, Principal Investigator — Tel-Aviv Sourasky Medical Center
Locations (1):
- Tel-Aviv Sourasky Medical Center, Tel Aviv, Israel